CLINICAL TRIAL: NCT01014676
Title: Probiotics and Infections in Children Attending Day Care Centres
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valio Ltd (Industry)
Collaborators: University of Helsinki (Other)
Other Study IDs: Valio-69
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Respiratory Tract Infections; Gastrointestinal Diseases
Keywords: Costs and Cost Analysis
MeSH Terms: conditions — Respiratory Tract Infections; Gastrointestinal Diseases | interventions — Probiotics

ARMS (2):
- Probiotic milk (Active Comparator)
  Interventions: Dietary Supplement: Probiotic
- Standard milk (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotic milk
Other: Placebo
  Arms: Standard milk

SUMMARY:
The purpose of this study is to evaluate the effect of regular consumption of probiotic milk in preventing illnesses in Finnish children attending day care centres, and possible cost-benefits that could be associated with fewer illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 6 years in the beginning of the intervention
* Attendance at a day care centre participating in the study (5 days a week)

Exclusion Criteria:

* Milk allergy or lactose intolerance
* Congenital heart diseases that requires regular medication
* Malign diseases
* Cytostatic treatment
* Use of biological rheumatic medication
* Continuous microbial medication
* Regular use of oral corticosteroids (inhalable accepted)
* Diabetes
* Simultaneous participation in other clinical trials

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Anne Pitkäranta, Professor, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Clinical Life Sciences Inc., Kajaani and Oulu, Province of Oulu, Finland

REFERENCES:
- [Derived] Korpela K, Salonen A, Virta LJ, Kumpu M, Kekkonen RA, de Vos WM. Lactobacillus rhamnosus GG Intake Modifies Preschool Children's Intestinal Microbiota, Alleviates Penicillin-Associated Changes, and Reduces Antibiotic Use. PLoS One. 2016 Apr 25;11(4):e0154012. doi: 10.1371/journal.pone.0154012. eCollection 2016. PMID 27111772